CLINICAL TRIAL: NCT06698419
Title: A Prospective Study: The Effect of RADA16 on Mastoid Cavity Epithelialization After Canal Wall Down Mastoidectomy
Brief Title: RADA16 on Mastoid Cavity Epithelialization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: 3-D Matrix UK Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202401064
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Delayed Wound Healing
Keywords: Mastoidectomy; Healing; Biologic; Mastoid cavity; Mastoid cavity disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the experimental group or the control group. All participants will undergo a canal wall down mastoidectomy in standard fashion. Participants in the experimental group will receive RADA16 gel in the mastoid cavity at the conclusion of the surgery whereas participants in the control group will not.
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeon/principal investigator performing the canal wall down mastoidectomy will be aware of participant allocation. Participants and research co-investigators will not be aware of patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RADA16 Group (Experimental): Participants will undergo canal wall down mastoidectomy in standard fashion. All participants will have absorbable gelatin sponge placed into the mastoid cavity which is standard care. Only participants in this arm will receive RADA16 gel into the mastoid cavity before placement of the gelatin sponge.
  Interventions: Device: RADA16 gel application into mastoid cavity
- Control Group (No Intervention): Participants will undergo canal wall down mastoidectomy in standard fashion. All participants will have absorbable gelatin sponge placed into the mastoid cavity which is standard care. Participants in this arm will not receive RADA16 gel.

INTERVENTIONS:
Device: RADA16 gel application into mastoid cavity — A single application of RADA16 gel will be applied along the surface of the mastoid cavity intraoperatively prior to insertion of gelatin sponge packing. Application will involve a thin layer of gel just enough to cover the entire surface of the cavity.
  Other Names: PuraGel
  Arms: RADA16 Group

SUMMARY:
The goal of this clinical trial is to see if the application of RADA16 gel can expedite and improve the healing process in participants after canal wall down mastoidectomy. The main questions are:

* Does application of RADA16 in the mastoid cavity after canal wall down mastoidectomy lead to faster healing (i.e. epithelialization)?
* Is application of RADA16 in the mastoid cavity after canal wall down mastoidectomy associated with a decreased need for medications after surgery (i.e. antibiotics, steroids), less frequent in-office debridements, and less postoperative appointments?

Researchers will compare the healing outcomes in participants treated with RADA16 gel to those in a control group who do not receive the treatment.

Participants will:

* Undergo canal wall down mastoidectomy as recommended regardless of participation in the clinical trial
* Follow-up postoperatively for clinical assessment at 1 month, 2 months, 3 months, 6 months, 1 year, 18 months, and 2 years. Participants may follow-up more frequently as needed.

DETAILED DESCRIPTION:
Canal wall-down mastoidectomy is a commonly performed procedure for the treatment of cholesteatoma and chronic otitis media which involves elimination of the posterior wall of the external auditory canal and creation of a mastoid cavity. Unlike its canal wall-up counterpart, canal wall-down mastoidectomy allows for exteriorization and removal of cholesteatoma and middle ear disease in otherwise difficult-to-access middle ear subsites (e.g., sinus tympani and lateral epitympanum), and improved surveillance of these spaces post-operatively.

While there are many benefits to canal wall-down mastoidectomy in the right patient, the creation of a mastoid cavity is not without pitfalls. Normally, the tympanic cavity and mastoid air cells are covered in mucosal epithelium which is important in middle ear ventilation, protection from infection, and sound transmission to the inner ear. A mastoid cavity requires life-long maintenance and care and periodic visits to an otolaryngologist for debridement and surveillance. In creation of the mastoid cavity, the mucosa lining tympanic cavity and mastoid air cells is often removed along with cholesteatoma or other middle ear disease leaving exposed bone. Maturation of the mastoid cavity requires re-epithelization of the cavity which can take months to years to occur [2]. Inadequate or delayed epithelialization results in an "unstable" mastoid cavity which occurs in 20 to 60% of patients depending on the study [2-4]. Formation of granulation tissue and adhesions trap debris and lead to excessive crusting, chronic otorrhea, and intolerance to water exposure which further hinders mastoid cavity healing. In the researchers' experience, these patients often require more frequent office visits for debridement, application of ototopical agents, in-office cauterization, and revision mastoidectomy under general anesthesia in some cases.

Creation of a mastoid cavity requires making a wide enough cavity to allow for adequate ventilation, facilitate cavity inspection, and promote a self-cleaning environment. Other anatomic factors important for the surgeon include creating a mastoid cavity that is oval-shaped with a low facial ridge [5]. Because maturation of the mastoid cavity requires complete epithelization, a variety of methods have been explored to facilitate this process including application of a gelatin film [6], silastic sheeting [7], pedicled postauricular periosteal flap [8], and poly-N-acetyl-glucosamine sheet with fibrin glue [9]. At our institution and many others, mastoid cavities are packed with absorbable gelatin sponge (Gelfoam) which provides structural support for the newly formed mastoid cavity by securing soft tissue and grafts in place.

To date, there are no studies evaluating the use of RADA16 gel in human otologic surgery. RADA16 is a viscous solution of synthetic peptides that self-assemble into a transparent hydrogel matrix at physiological pH, mimicking the native extracellular matrix [10]. This unique property has enabled RADA16 to be adapted for various clinical applications. The biologic scaffold created by RADA16 acts as a physical barrier over wounds, inhibiting blood flow and promoting hemostasis. Its effectiveness has been demonstrated in various cardiovascular, gastrointestinal, and otolaryngologic procedures specifically endonasal [11-17].

The hydrogel matrix of RADA16 not only serves as a barrier but also acts as a biologic scaffold that supports wound healing, cell proliferation, and tissue regeneration [18]. Numerous in vivo studies have highlighted RADA16's potential as a wound healing agent. For example, it has shown promise in promoting mucosal regeneration after gastric ulcer formation [19], colon injury in a rat model [20], periodontal disease [21], and following endoscopic excision of gastrointestinal lesions [17]. Animal models have also demonstrated RADA16's ability to prevent scarring and adhesion formation, specifically in preventing esophageal stricture after submucosal resection [22]. In sinonasal surgery, RADA16 has proven beneficial in enhancing wound healing, preventing adhesion formation, and minimizing crusting [13, 23]. In a sheep model, RADA16 application to nasal mucosal defects led to reduced adhesion formation and accelerated healing [24]. More pertinent to this investigation, a study using a middle ear rodent model revealed that cultured middle ear epithelial cells treated with RADA16 were able to survive and repair mucosal defects, unlike those not treated with RADA16 [25].

Given the previous studies which include improved mucosal wound healing in the sinonasal cavity and a promising middle ear rodent study, researchers' aim to investigate and compare mastoid cavity epithelization rates after canal wall down mastoidectomy with and without the intraoperative application of RADA16 gel.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults over the age of 18 years who require a canal wall down mastoidectomy for any reason including cholesteatoma, chronic suppurative middle ear disease, and neoplasm.
* Participants with history of canal wall up mastoidectomy who now require canal wall down mastoidectomy for any reason.

Exclusion Criteria:

* History of chronic immunodeficiency and autoimmune disease
* History of head and neck radiation
* Active tobacco use
* History of coronary artery disease
* History of peripheral vascular disease
* History of diabetes mellitus
* Known allergy to RADA16 gel or its components
* Vulnerable populations including children, neonates, pregnant women, prisoners, institutionalized individuals, and other individuals who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to Complete Mastoid Cavity Epithelialization at 1 Month | Baseline and Postoperative Month 1
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 2 Months | Baseline and Postoperative Month 2
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 3 Months | Baseline and Postoperative Month 3
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 6 Months | Baseline and Postoperative Month 6
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 1 Year | Baseline and Postoperative Year 1
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 18 Months | Baseline and Postoperative Month 18
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.
Time to Complete Mastoid Cavity Epithelialization at 2 Years | Baseline and Postoperative Year 2
  The mastoid cavity will be evaluated postoperatively using an operative microscope. The principal investigator will record the otoscopic exam which will be saved as a digital file on a password-secured server. Two separate investigators who are masked to participant arm allocation will view the recorded exam and evaluate the mastoid cavity for complete epithelialization.

SECONDARY OUTCOMES:
Total Number of Medications Prescribed Up To Complete Epithelialization | Baseline to complete epithelialization, up to 2 years
  The total number of medications prescribed postoperatively to promote mastoid cavity healing will be assessed with focus on antibiotics and steroids.
Total Number of Mastoid Cavity Debridements Up to Complete Epithelialization | Baseline to complete epithelialization, up to 2 years
  The total number of in-office mastoid cavity debridements will be recorded and assessed. Participants with faster and more robust healing are expected to require less in-office debridements.
Total Number of Postoperative Visits Up to Complete Epithelialization | Baseline to complete epithelialization, up to 2 years
  The total number of postoperative visits (including set time points at 1 month, 2 months, 3 months, 9 months, 1 year, 18 months, and 2 years) will be recorded and assessed. Participants with faster and more robust healing are expected to not need additional visits, specifically for mastoid cavity healing related problems.

CONTACTS AND LOCATIONS:
Overall Officials: Rex Haberman, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD with other researchers.

REFERENCES:
- [Background] Akiyama N, Yamamoto-Fukuda T, Takahashi H, Koji T. In situ tissue engineering with synthetic self-assembling peptide nanofiber scaffolds, PuraMatrix, for mucosal regeneration in the rat middle-ear. Int J Nanomedicine. 2013;8:2629-40. doi: 10.2147/IJN.S47279. Epub 2013 Jul 24. PMID 23926427
- [Background] Lee MF, Ananda A. Self-assembling RADA16 peptide hydrogel supports hemostasis, synechiae reduction, and wound healing in a sheep model of endoscopic nasal surgery. Auris Nasus Larynx. 2023 Jun;50(3):365-373. doi: 10.1016/j.anl.2022.09.012. Epub 2022 Oct 22. PMID 36283900
- [Background] Friedland Y, Bagot d'Arc MBD, Ha J, Delin C. The Use of Self-Assembling Peptides (PuraStat) in Functional Endoscopic Sinus Surgery for Haemostasis and Reducing Adhesion Formation. A Case Series of 94 Patients. Surg Technol Int. 2022 Nov 15;41:105-110. doi: 10.52198/22.STI.41.GS1694. PMID 35556241
- [Background] Oumrani S, Barret M, Bordacahar B, Beuvon F, Hochart G, Pagnon-Minot A, Coriat R, Batteux F, Prat F. Application of a self-assembling peptide matrix prevents esophageal stricture after circumferential endoscopic submucosal dissection in a pig model. PLoS One. 2019 Mar 12;14(3):e0212362. doi: 10.1371/journal.pone.0212362. eCollection 2019. PMID 30861007
- [Background] Takeuchi T, Bizenjima T, Ishii Y, Imamura K, Suzuki E, Seshima F, Saito A. Enhanced healing of surgical periodontal defects in rats following application of a self-assembling peptide nanofibre hydrogel. J Clin Periodontol. 2016 Mar;43(3):279-88. doi: 10.1111/jcpe.12515. Epub 2016 Mar 2. PMID 26788695
- [Background] Araki T, Mitsuyama K, Yamasaki H, Morita M, Tsuruta K, Mori A, Yoshimura T, Fukunaga S, Kuwaki K, Yoshioka S, Takedatsu H, Kakuma T, Akiba J, Torimura T. Therapeutic Potential of a Self-Assembling Peptide Hydrogel to Treat Colonic Injuries Associated with Inflammatory Bowel Disease. J Crohns Colitis. 2021 Sep 25;15(9):1517-1527. doi: 10.1093/ecco-jcc/jjab033. PMID 33596312
- [Background] Kakiuchi Y, Hirohashi N, Murakami-Murofushi K. The macroscopic structure of RADA16 peptide hydrogel stimulates monocyte/macrophage differentiation in HL60 cells via cholesterol synthesis. Biochem Biophys Res Commun. 2013 Apr 12;433(3):298-304. doi: 10.1016/j.bbrc.2013.02.105. Epub 2013 Mar 19. PMID 23518074
- [Background] Uraoka T, Ochiai Y, Fujimoto A, Goto O, Kawahara Y, Kobayashi N, Kanai T, Matsuda S, Kitagawa Y, Yahagi N. A novel fully synthetic and self-assembled peptide solution for endoscopic submucosal dissection-induced ulcer in the stomach. Gastrointest Endosc. 2016 Jun;83(6):1259-64. doi: 10.1016/j.gie.2015.11.015. Epub 2015 Dec 1. PMID 26608126
- [Background] Subramaniam S, Kandiah K, Chedgy F, Fogg C, Thayalasekaran S, Alkandari A, Baker-Moffatt M, Dash J, Lyons-Amos M, Longcroft-Wheaton G, Brown J, Bhandari P. A novel self-assembling peptide for hemostasis during endoscopic submucosal dissection: a randomized controlled trial. Endoscopy. 2021 Jan;53(1):27-35. doi: 10.1055/a-1198-0558. Epub 2020 Jul 17. PMID 32679602
- [Background] Stenson KM, Loftus IM, Chetter I, Fourneau I, Cavanagh S, Bicknell C, Loftus P. A Multi-Centre, Single-Arm Clinical Study to Confirm Safety and Performance of PuraStat(R), for the Management of Bleeding in Elective Carotid Artery Surgery. Clin Appl Thromb Hemost. 2022 Jan-Dec;28:10760296221144307. doi: 10.1177/10760296221144307. PMID 36514251
- [Background] Pioche M, Camus M, Rivory J, Leblanc S, Lienhart I, Barret M, Chaussade S, Saurin JC, Prat F, Ponchon T. A self-assembling matrix-forming gel can be easily and safely applied to prevent delayed bleeding after endoscopic resections. Endosc Int Open. 2016 Apr;4(4):E415-9. doi: 10.1055/s-0042-102879. Epub 2016 Mar 30. PMID 27092320
- [Background] Morshuis, M., M. Schönbrodt, and J. Gummert, Safety and Performance of a Self-Assembling Peptide Haemostat for the Management of Bleeding after Left Ventricular Assist Device Implantation: Outcomes of a Post Market Clinical Follow-Up Study. Journal of Heart and Lung Transplantation, 2019. 38(4): p. S194-S194.
- [Background] Lee MF, Ma Z, Ananda A. A novel haemostatic agent based on self-assembling peptides in the setting of nasal endoscopic surgery, a case series. Int J Surg Case Rep. 2017 Nov 20;41:461-464. doi: 10.1016/j.ijscr.2017.11.024. eCollection 2017. PMID 29546017
- [Background] Giritharan S, Salhiyyah K, Tsang GM, Ohri SK. Feasibility of a novel, synthetic, self-assembling peptide for suture-line haemostasis in cardiac surgery. J Cardiothorac Surg. 2018 Jun 15;13(1):68. doi: 10.1186/s13019-018-0745-2. PMID 29903028
- [Background] Branchi F, Klingenberg-Noftz R, Friedrich K, Burgel N, Daum S, Buchkremer J, Sonnenberg E, Schumann M, Treese C, Troger H, Lissner D, Epple HJ, Siegmund B, Stroux A, Adler A, Veltzke-Schlieker W, Autenrieth D, Leonhardt S, Fischer A, Jurgensen C, Pape UF, Wiedenmann B, Moschler O, Schreiner M, Strowski MZ, Hempel V, Huber Y, Neumann H, Bojarski C. PuraStat in gastrointestinal bleeding: results of a prospective multicentre observational pilot study. Surg Endosc. 2022 May;36(5):2954-2961. doi: 10.1007/s00464-021-08589-6. Epub 2021 Jun 15. PMID 34129089
- [Background] Sankar S, O'Neill K, Bagot D'Arc M, Rebeca F, Buffier M, Aleksi E, Fan M, Matsuda N, Gil ES, Spirio L. Clinical Use of the Self-Assembling Peptide RADA16: A Review of Current and Future Trends in Biomedicine. Front Bioeng Biotechnol. 2021 Jun 2;9:679525. doi: 10.3389/fbioe.2021.679525. eCollection 2021. PMID 34164387
- [Background] Kobayashi T, Gyo K, Komori M, Hyodo M. Polyglycolic acid sheet attached with fibrin glue can facilitate faster epithelialization of the mastoid cavity after canal wall-down tympanoplasty. Auris Nasus Larynx. 2017 Dec;44(6):685-689. doi: 10.1016/j.anl.2017.01.013. Epub 2017 Feb 20. PMID 28215637
- [Background] Kanemaru S, Hiraumi H, Omori K, Takahashi H, Ito J. An early mastoid cavity epithelialization technique using a postauricular pedicle periosteal flap for canal wall-down tympanomastoidectomy. Acta Otolaryngol Suppl. 2010 Nov;(563):20-3. doi: 10.3109/00016489.2010.496463. PMID 20879813
- [Background] Ng M, Linthicum FH Jr. Long-term effects of Silastic sheeting in the middle ear. Laryngoscope. 1992 Oct;102(10):1097-102. doi: 10.1288/00005537-199210000-00002. PMID 1328786
- [Background] McGhee MA, Dornhoffer JL. The effect of gelfilm in the prevention of fibrosis in the middle ear of the animal model. Am J Otol. 1999 Nov;20(6):712-6. PMID 10565713
- [Background] Wormald PJ, Nilssen EL. The facial ridge and the discharging mastoid cavity. Laryngoscope. 1998 Jan;108(1 Pt 1):92-6. doi: 10.1097/00005537-199801000-00017. PMID 9432074
- [Background] Henatsch D, Alsulami S, Duijvestijn AM, Cleutjens JP, Peutz-Kootstra CJ, Stokroos RJ. Histopathological and Inflammatory Features of Chronically Discharging Open Mastoid Cavities: Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Mar 1;144(3):211-217. doi: 10.1001/jamaoto.2017.2801. PMID 29327047
- [Background] Beales PH. Complications following obliterative mastoid operations. Arch Otolaryngol. 1969 Jan;89(1):196-8. doi: 10.1001/archotol.1969.00770020198035. No abstract available. PMID 4882186
- [Background] Thiel G, Rutka JA, Pothier DD. The behavior of mastoidectomy cavities following modified radical mastoidectomy. Laryngoscope. 2014 Oct;124(10):2380-5. doi: 10.1002/lary.24610. Epub 2014 Jul 14. PMID 24459037
- [Background] Kerckhoffs KG, Kommer MB, van Strien TH, Visscher SJ, Bruijnzeel H, Smit AL, Grolman W. The disease recurrence rate after the canal wall up or canal wall down technique in adults. Laryngoscope. 2016 Apr;126(4):980-7. doi: 10.1002/lary.25591. Epub 2015 Sep 25. PMID 26404516